CLINICAL TRIAL: NCT05477888
Title: Psychometric Properties of the Chinese Version of Penn State [Electronic] Cigarette Dependence Index
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, A.P., Sun Yat-sen University
Other Study IDs: wjn-ChiCTR2200060896
Record Dates: First submitted 2022-07-24; First posted 2022-07-28 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: E-Cig Use
Keywords: Adolescent; Electronic Nicotine Delivery Systems / psychology; Psychometrics
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urinal cotinine and exhaled carbon monoxide
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaires assessed e-cigarette users: 1. ≥18 years old;
  2. Those who used e-cigarettes at least once a week for the past month;
  3. Be able to read and communicate in Chinese.
  Interventions: Other: Questionnaires set

INTERVENTIONS:
Other: Questionnaires set — Participants will be asked to respond to the demographic information sheet,e-cigarette using characteristics sheet,the Penn State Electronic Cigarette Dependence Index (PS-ECDI ).

SUMMARY:
The purpose of this study is to realize the first evaluation of the psychometric characteristics of the Chinese version of the the Penn State University Electronic Cigarette Dependence Index Scale.

DETAILED DESCRIPTION:
This study will use forward translation, reverse translation, and comprehensive methods to Chinese-translate the Penn State University Electronic Cigarette Dependence Index Scale to form a Chinese version of the Penn State University Electronic Cigarette Dependence Index Scale that is more in line with the Chinese language and cultural environment. This study will also verify its reliability and validity in a large sample population to form a formal version of the scale. The scale will provide an effective tool for evaluating the degree of e-cigarette dependence among young people and adolescents in my country.

ELIGIBILITY:
Inclusion Criteria:

* (1)≥18 years old;
* (2)Those who used e-cigarettes at least once a week for the past month;
* (3)Be able to read and communicate in Chinese.

Exclusion Criteria:

* Those who are unable to communicate due to serious mental or physical illnesses such as deafness, confusion caused by mental illness, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total number of 275 adults who used nicotine-containing e-cigarettes at least once a week for the past month and have smoked daily for the last 3 months
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
E-cigarette dependence | Baseline
  The Penn State Electronic Cigarette Dependence Index is a validated self-reported instrument assessing e-cigarette dependence.Possible scales range from 0(no dependence) to 20(high dependency).

SECONDARY OUTCOMES:
Self-reported addiction | Baseline
  Measured by a 0-100 point scale：the higher the score of the participant, the more severe the dependence on e-cigarettes.
Time to first vape | Baseline
  Corroborative evidence for e-cigarette dependence：the shorter the time interval, the greater the dependence on e-cigarettes.
Vapes/day and vaping days/week | Baseline
  Corroborative evidence for e-cigarette dependence：the higher the frequency, the more severe the dependence on e-cigarettes.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- XIAW, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The non-identified individual participant data will be shared after the outcomes have been published.
Supporting Information: SAP
Time Frame: After the publication of the study.
Access Criteria: Researchers should contact the PI for approval of the study protocol.